CLINICAL TRIAL: NCT01311037
Title: The Combination of GnRh Analogue and Aromatase Inhibitor in Receptor Positive Premenopausal Women With Advanced Breast Cancer A Prospective Trial
Brief Title: The Combination of GnRh Analogue and Aromatase Inhibitor in Receptor Positive Premenopausal Women With Advanced Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2081-064; RAC# 2081-064
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Advanced Breast Cancer
Keywords: Premenopausal Women with Advanced Breast Cancer
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: GnRh Analogue and Aromatase Inhibitor — GnRh Analogue and Aromatase Inhibitor

SUMMARY:
The Combination of GnRh Analogue and Aromatase Inhibitor in Receptor Positive Premenopausal Women with Advanced Breast Cancer A Prospective Trial.

DETAILED DESCRIPTION:
The Combination of GnRh Analogue and Aromatase Inhibitor in Receptor Positive Premenopausal Women with Advanced Breast Cancer A Prospective Trial.

ELIGIBILITY:
Inclusion Criteria:

* Receptor Positive Premenopausal Women with Advanced Breast Cancer.

Exclusion Criteria:

* Any woman other than diagnosis of Receptor Positive Premenopausal with Advanced Breast Cancer.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Receptor Positive Premenopausal Women with Advanced Breast Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2009-01

CONTACTS AND LOCATIONS:
Overall Officials: Al Sayed, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia